CLINICAL TRIAL: NCT01157611
Title: The Effect of Online Based Mentoring Program on the Blood Glucose and Satisfaction Score in Type 1 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jae Hyeon Kim, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-05-065
Record Dates: First submitted 2010-07-05; First posted 2010-07-07 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Type 1 Diabetes
Keywords: online based mentoring program,; type 1 diabetes,; blood glucose,; satisfaction score
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mentoring program group (Active Comparator): type 1 diabetes patients participating in online base mentoring program
  Interventions: Behavioral: Mentoring program
- Control group (No Intervention): type 1 diabetes patients receiving regular clinic visits

INTERVENTIONS:
Behavioral: Mentoring program — mentoring program group patients should register their SMBG, exercise, food intake and insulin dose on the website designed for this study and receive advices of mentors from peer group.
  Other Names: online based mentoring program
  Arms: Mentoring program group

SUMMARY:
Purpose:

To evaluate the effects of online based mentoring program on the blood glucose and satisfaction score in type 1 diabetes patients. Peer group mentoring will be as effective as guidance by the doctors.

Methods:

80 type 1 patients will be randomly divided into two groups (e.g. mentoring program group and control group). All patients will receive routine check up and blood test for ordinary type 1 patients. In addition, program group patients should register their SMBG, exercise, food intake and insulin dose on the website designed for this study and receive advices of mentors from peer group. Every patient will submit questionnaire on the first day of the study and the last day(after 12 weeks) of the study.

DETAILED DESCRIPTION:
Subjects with T1DM on intensive insulin therapy and with hemoglobin A1c (HbA1c) ≥8.0% were randomized to mentored (glucometer transmission with feedback from mentors) or control (glucometer transmission without feedback) groups and were examined for 12 weeks. Five mentors were interviewed and selected, of which two were T1DM patients themselves and three were parents with at least one child diagnosed with T1DM since more than 5 years ago.

ELIGIBILITY:
Inclusion Criteria:

* age > 18, more than 6 month after the diagnosis of type 1 diabetes
* HbA1c > 8% despite of multiple insulin injection or insulin pump
* who are capable of using the internet

Exclusion Criteria:

* pregnant women
* who cannot use the internet
* those who does not want to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
change of the blood glucose | week 0 (baseline), 6, 12
  HbA1c, Fructosamine

SECONDARY OUTCOMES:
satisfaction score | week 0 (baseline), 6, 12
  incidence of hypoglycemia, numbers of daily SMBG, DTSQs, DTSQc, ADDQoL

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hyeon Kim, M.D., Ph. D., Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea